CLINICAL TRIAL: NCT05166564
Title: A Randomised Controlled Trial to Evaluate the Effect of a Protein Enriched Mediterranean Diet and Exercise Intervention on the Nutritional Status and Cognitive Performance of Adults At Risk of Undernutrition and Cognitive Decline
Brief Title: The PROtein Enriched MEDiterranean Diet and EXercise Trial for Older Adults At Risk of Undernutrition
Acronym: PROMED-EX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: University College Dublin (Other); Wageningen University (Other); Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); Dublin City University (Other)
Responsible Party: Principal Investigator, Claire McEvoy, PROMED-EX Principal Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B21/16; BB/V019201/1 (Other Grant/Funding Number: European Joint Programming Initiative (HDHL)); BB/V019201/1 (Other Grant/Funding Number: UK Research & Innovation (UKRI):BBSRC MRC)
Record Dates: First submitted 2021-09-17; First posted 2021-12-22 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Impairment; Poor Nutrition; Cognitive Decline
Keywords: Poor nutrition; Older adults; Cognitive impairment; Cognitive decline; Mediterranean Diet; Protein enriched Mediterranean Diet
MeSH Terms: conditions — Cognitive Dysfunction; Malnutrition | interventions — Methods; Exercise

STUDY DESIGN:
Intervention Model Description: This study is a single blind parallel randomised controlled trial design, recruiting n=105 eligible participants and randomising into one of three groups with n=35 participants assigned into each group. Group 1: a Protein enriched Mediterranean diet (PROMED) Intervention; Group 2: a Protein enriched Mediterranean diet and exercise (PROMED-EX) intervention; and Group 3: the control group. The active intervention arms will last for three months with an additional three months of follow-up. Data will be collected from participants at study baseline, 3months and 6 months. The study statistician - independent of study recruitment, intervention delivery and data collection - has generated the randomisation scheme using a computer generated random number sequence (Release 14 StataCorp LP, College Station) assigning participant ID numbers to either the PROMED, the PROMED-EX or the control group using block randomisation in blocks of 6.
Who Masked: Outcomes Assessor
Masking Description: Sealed opaque envelopes have been prepared by a member of the research team (independent of data collection). Envelops numbered with study IDs will conceal the allocated group assignment from the research team involved in screening and recruitment. Participants will be allocated a study ID number at baseline once written consent to participate has been provided. After completion of baseline measurements, a researcher (independent of outcome measurements) will open the sealed envelope corresponding to the participant's study ID to reveal the allocated group and arrange intervention delivery if required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PROMED (Experimental Intervention 1) (Experimental): A Protein Enriched Mediterranean Diet (PROMED) intervention. Participants will receive individually tailored resources to encourage adoption of a protein-enriched Mediterranean diet pattern.
  Interventions: Behavioral: A Protein Enriched Mediterranean Diet (PROMED) Intervention
- PROMED-EX (Experimental Intervention 2) (Experimental): A Protein Enriched Mediterranean Diet & Exercise (PROMED-EX) Intervention. Participants will receive the same PROMED diet resources (Experimental Intervention 1) and an individually tailored exercise intervention.
  Interventions: Behavioral: A Protein Enriched Mediterranean Diet & Exercise (PROMED-EX) Intervention
- Control group (No Intervention): 'Standard Care' - consisting of a general diet information sheet.

INTERVENTIONS:
Behavioral: A Protein Enriched Mediterranean Diet (PROMED) Intervention — Researchers will provide individually tailored dietary advice and written materials to encourage 'a little and often' meal plan to support adoption of the PROMED intervention. The daily energy and protein requirements of each participant will be calculated based on National Institute of Health & Care Excellence guidance for Nutrition Support in Adults at Risk of Malnutrition. Several resources have been developed to facilitate behaviour change: a) A PROMED Diet Information Booklet to include an overview of the PROMED Diet, tips for incorporating more PROMED foods into the diet and information on the health benefits of a PROMED diet, b) A PROMED Recipe Book offering ideas for breakfast, lunch and dinner as well as suitable snack ideas and c) key PROMED foods ordered through a local supermarket's online delivery service and delivered to participants' homes on a weekly or fortnightly basis for the 3-month active intervention phase.
  Arms: PROMED (Experimental Intervention 1)
Behavioral: A Protein Enriched Mediterranean Diet & Exercise (PROMED-EX) Intervention — Participants will receive a dietary intervention identical to PROMED participants, plus an exercise intervention. The home-based exercises are based on a modified version of the 'ExWell@home' programme developed by health professionals with significant expertise in community-based exercise rehabilitation for chronic disease. Cardiorespiratory fitness will be determined using a 3-minute step test and pulse rate. Participants will receive access to pre-recorded exercise classes and a written resource designed for older adults (ExWell@home) and adapted for the current study. Participants will be encouraged to complete two sessions per week (30-60 minutes per session). To cater for differing abilities, four levels of classes will be available for participants: Chair based, basic, standard and advanced.
  Arms: PROMED-EX (Experimental Intervention 2)

SUMMARY:
PROMED-EX is a single-blind, parallel group randomised controlled trial to determine the effect of a PROtein enriched MEDiterranean diet (PROMED) in comparison to a PROtein enriched MEDiterranean diet and EXercise (PROMED-EX) intervention, or standard care on the nutritional status and cognitive performance of older undernourished adults with subjective cognitive decline.

DETAILED DESCRIPTION:
Undernutrition is common in older adults and can cause significant negative impacts on the health of older people, leading to weight loss and decline in cognitive function (memory and thinking abilities), loss of independence and hospitalisation. Undernutrition is associated with £23.5 billion/year in health and social care costs in the United Kingdom - over half of these costs are related to undernutrition in older adults.

Research suggests that undernutrition and weight loss occur a long time (at least 10 years) before the symptoms of cognitive decline become apparent. This means that correcting undernutrition and weight loss could help to prevent the onset of cognitive impairment.

The aim of the PROMED-EX trial is to test the effect of a 6-month protein enriched Mediterranean diet, with and without exercise, on the risk of undernutrition and cognitive decline in older adults in Northern Ireland. The PROMED-EX trial will recruit 105 older adults living in the community, at risk of poor nutrition, with a decline in memory but without a diagnosed cognitive impairment. Investigators will collect several measurements to determine the nutritional status and cognitive functioning of study participants and will repeat measurements during the study (at the start of the study, at 3 months (study midpoint) and at 6 months (study endpoint).

The goal is to identify potential effective solutions to undernutrition which can reduce cognitive decline and other negative health impacts on older adults. The research can be used to guide public health dietary guidelines for older people to prevent undernutrition and increase healthy life years.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling (non-institutionalised) participants ≥60 years older
* A high risk of undernutrition as defined by a Mini Nutritional Assessment -Short Form (MNA-SF) score of 8 - 11
* Positive screen for Subjective Cognitive Decline (SCD)

Exclusion Criteria:

* Cognitive impairment determined by the Mini Mental State Assessment (MMSE) or Telephone Cognitive Screen (T-CogS)
* Receiving oral or artificial nutritional support or medical food supplements
* Taking high dose nutritional supplements (supplements above the Reference Nutrient Intake levels).
* Dietary restrictions/allergies that limit ability to adhere to study requirements
* A diagnosis of mild cognitive impairment or dementia
* Dysphagia
* Chronic kidney disease
* Poorly controlled diabetes (HbA1c >8% or diabetes complications)
* Severe visual or language impairment
* Self-reported psychiatric problems or significant medical co-morbidities that compromise the ability to take part/limit capacity to consent
* Diagnosis of a comorbid condition that may alter performance on cognitive tests, e.g. stroke, head injury, Parkinson's disease, learning disabilities.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Mini Nutritional Assessment Score- Long Form | Baseline and 6 months
  The Primary outcome is change at 6 months (study endpoint) in Mini Nutritional Assessment (MNA) score between the two intervention groups and the control group. The MNA is a well validated tool with good sensitivity and specificity for predicting nutritional risk in older community dwelling adults. Scores range from 0-30 with a lower score reflecting poorer nutritional status.

SECONDARY OUTCOMES:
Mini Nutritional Assessment Score (midpoint change) | Baseline and 3 months
  Change at 3 months from baseline in Mini Nutritional Assessment (MNA) score between the two intervention groups and the control group. The MNA is a well validated tool with good sensitivity and specificity for predicting nutritional risk in older community dwelling adults. Scores range from 0-30 with a lower score reflecting poorer nutritional status.
Nutrient intake: PROMED Mediterranean Diet Score | Baseline, 3 months and 6 months
  Change at 3 and 6 months in Mediterranean Diet Score (MDS)(score range 0-14) between the two intervention groups and control. Higher scores reflect greater adherence to a Mediterranean diet.
Nutrient intake: (4 day food diary) | Baseline, 3 months and 6 months
  Change at 3 and 6 months in nutrient intakes (including protein intake) between the two intervention groups and control.
Simplified Nutrition Appetite Questionnaire (SNAQ) | Baseline, 3 months and 6 months
  Change in appetite at 3 and 6 months (from baseline). This is a brief 4-item questionnaire (score range 0-4) with lower scores suggesting deterioration of appetite.
Body Water (%) | Baseline, 3 months and 6 months
  Change in Body water (%) at 3 and 6 months (from baseline) using Bioelectrical Impedance Analysis (BodyStat 1500)
Total Body Fat (%) | Baseline, 3 months and 6 months
  Change in Total Body Fat (%) at 3 and 6 months (from baseline) using Bioelectrical Impedance Analysis (BodyStat 1500)
Lean Muscle Mass (kg) | Baseline, 3 months and 6 months
  Change in Muscle Mass (kg) at 3 and 6 months (from baseline) using Bioelectrical Impedance Analysis (BodyStat 1500)
Weight (kg) and height (cm) | Baseline, 3 months and 6 months
  Change in weight (kg) and Height (cm) at 3 and 6 months (from baseline). Both measurements will be used to calculate change in Body Mass Index (BMI) (Kg/m^2) across groups at 3 and 6 months.
Waist circumference (cm) | Baseline, 3 months and 6 months
  Change in waist circumference at 3 and 6 months (from baseline)
Physical Activity determined by completion of a Recent Physical Activity Questionnaire | Baseline, 3 months and 6 months
  Change at 3 and 6 months (from Baseline) in physical activity levels between the two intervention groups and control. This questionnaire inquires about physical activity across four domains (leisure time, occupation, commuting, and domestic life) during the past 4 weeks. Metabolic Equivalent of Task scores can be calculated and an estimation of total energy expenditure across the four domains.
Capturing Changes in Cognition (Catch-Cog) | Baseline, 3 months and 6 months
  Change at 3 and 6 months (from baseline) in cognition using the Capturing Changes in Cognition- Catch-Cog score. This composite includes an Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) word recognition (Sub score 0-12), ADAS-Cog orientation (Sub score 0-8), Controlled Oral Word Association Test (COWAT) (max number of words in 1 minute), Category Fluency Test (max number of words in 1 minute), a Digital Symbol Substitution test (correct number of symbols matched in 90 seconds), and an ADAS-Cog Word Recall Test (sub score range: 0-10). A higher score reflects better cognitive performance.
Trail Making Tests (TMT) (Part A & B) | Baseline, 3 months and 6 months
  Change in completion time of the TMT at 3 and 6 months (from baseline). Higher time reflects greater impairment.
Delayed recall test (0-10) | Baseline, 3 months and 6 months
  Change at 3 and 6 months (from baseline) in a delayed recall test of recalled learned words after a 5-minute delay (score range 0-10)
Functional performance measured using the Short Physical Performance Battery (SPPB) test. | Baseline, 3 months and 6 months
  Change at 3 and 6 months in functional performance from baseline (using the SBBP): The SPPB will test participant's Gait (time to walk 8 feet), Balance (ability to complete a side-by-side, a semi-tandem and a tandem stand) and Strength (time to complete 5 chair stands). Category scores range from 0-4 and total score (0-12) with a higher score representing better physical functioning.
Grip Strength measured by isometric grip force (0-100kg) | Baseline, 3 months and 6 months
  Change in isometric grip force (0-100kg) at 3 and 6 months (from baseline) using a Dynamometer
Health-related quality of life (Short Form (SF)-36) | Baseline, 3 months and 6 months
  Change in health related quality of life measures at 3 and 6 months between the two intervention groups and control. The SF-36 is a 36-item questionnaire (covering 8 domains of health including physical functioning; role limitations due to physical health; role limitation due to emotional problems; energy/fatigue; emotional well-being; social functioning; pain; general health.Scores range from 0-100 with higher score indicating a better quality of life.
Geriatric Depression Scale | Baseline, 3 months and 6 months
  Change in Depression scale at 3 and 6 months (from baseline) Scores range from 0-15. A score ≥5 indicates probable depression
Systolic Blood Pressure (mmHg) | Baseline, 3 months and 6 months
  Change at 3 and 6 months (from baseline) using a Omron automated blood pressure monitor
Diastolic Blood Pressure (mmHg) | Baseline, 3 months and 6 months
  Change at 3 and 6 months (from baseline) using an Omron automated blood pressure monitor
Biochemical markers: nutritional, cardiometabolic and inflammatory | Baseline, 3 months and 6 months
  Blood sample will be collected to determine change in serum levels of Vitamin A, Vitamin E , Carotenoids (nmol/l), change in serum lipid profile (Total cholesterol, HDL cholesterol, LDL Cholesterol and triglycerides (mmol/l)), HbA1c (mmol/mol) , fasting plasma glucose (mmol/l) and Insulin (pmol/l), High Sensitivity C-Reactive Protein (mg/l), Interleukin-6 (pg/ml),at 3 and 6 months (from Baseline).

OTHER OUTCOMES:
Explore the acceptability and tolerance of the intervention | 6 months
  A study evaluation questionnaire will be administered to participants at 6 months to determine acceptability, tolerance and potential adverse effects of the intervention components and the intervention materials
Exploratory outcome: Metabolomic profiling | Baseline, 3 months and 6 months
  The blood samples required for Metabolomics analysis will be transferred to University College Dublin.
  An exploratory outcome using both targeted and untargeted approaches. Metabolomics will be performed using NMR and LC-MS-based approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Claire McEvoy, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queen's University Belfast, Belfast, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited in free open access repositories e.g. Queen's University Belfast (QUB) Pure Research portal and Zenodo (https://zenodo.org/), with guaranteed preservation of for ten years or more in order to maximise discovery and data sharing opportunities. The study description and variable metadata catalogues will be published also. Where possible, metadata will be made available through the Joint Programme Initiative: a Healthy Diet for a Healthy Life (JPI-HDHL) Meta Database (http://www.jpihdhl.eu) to maximise the visibility to the wider research community.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available once statistical analyses have been complete and for 10 years thereafter.
Access Criteria: The following conditions will apply to data use:
  * agreement on methodology
  * allowance to link the dataset with other datasets
  * data security
  * agreement on publication and authorship

REFERENCES:
- [Derived] Ward NA, Reid-McCann R, Brennan L, Cardwell CR, de Groot C, Maggi S, McCaffrey N, McGuinness B, McKinley MC, Noale M, O'Neill RF, Prinelli F, Sergi G, Trevisan C, Volkert D, Woodside JV, McEvoy CT. Effects of PROtein enriched MEDiterranean Diet and EXercise on nutritional status and cognition in adults at risk of undernutrition and cognitive decline: the PROMED-EX Randomised Controlled Trial. BMJ Open. 2023 Oct 25;13(10):e070689. doi: 10.1136/bmjopen-2022-070689. PMID 37880167
- See also: Link to PROMED-COG consortium and trial website — https://www.qub.ac.uk/sites/promed-cog/